CLINICAL TRIAL: NCT05307081
Title: A Prospective, Observational, Consecutive, Qualitative, Multicenter Study Assessing Eye Drop Administration
Brief Title: An Observational, Qualitative Study Assessing Eye Drop Administration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TEAR-2020-401
Record Dates: First submitted 2020-10-22; First posted 2022-04-01 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Ocular Injury
MeSH Terms: conditions — Eye Injuries | interventions — Lubricant Eye Drops

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: Artificial Tears

INTERVENTIONS:
Drug: Artificial Tears — Artificial Tears are an FDA approved intervention

SUMMARY:
This is a prospective, observational, consecutive, qualitative, multicenter study. Based on the available published evidence that supports patient challenges with eyedrop administration, the purpose of this video-capture study is to evaluate a more real-world population of consenting patients, regardless of age, with or without visual impairment, at routine eyecare visits.

To date, no studies have been performed evaluating a real-world population consisting of daily routine eyecare clinic patients with or without visual impairment. This study will help to determine the ability to achieve success with self-administration of eyedrops in the real world.

DETAILED DESCRIPTION:
Introduction: This is a prospective, observational, consecutive, qualitative, multicenter study. A robust body of evidence suggests patients demonstrate challenges with eyedrop adherence and improper administration. The current standard of care following ophthalmic surgery is topical treatment with corticosteroids, antibiotics, and NSAIDs. Prospectively evaluated patients accuracy in administering eyedrops, during the post-operative period of cataract surgery, with 92.6% of patients demonstrating at least one type of improper administration technique. Few examples of possible errors included neglect of handwashing, failure to shake the eyedrop bottle, contamination of the bottle tip, incorrect amount of drops, and even missing the ocular surface entirely. Additionally, there was an incongruence between patient's impression of their technique and physician's observation. Thirty-five percent of patients who reported not missing the eye, did miss the eye under observation, and 39.3% of the patients who believed they never touched the eye with the bottle tip, did touch the ocular surface.

Similar studies were also performed in visually impaired patients due to glaucoma and retinal diseases with up to 47% of patients with retinal diseases touching the bottle to the eye, and up to 30% of patients not being able to administer a drop into the eye.

The objective of this study is to assess the accuracy of successful eye drop administration in patients undergoing routine exams.

This study also seeks to understand the discrepancy between patient impressions of eyedrop instillation success compared to success determined by ophthalmologist and optometrist evaluation.

Study Design This study will video capture adult subjects or Legal Authorized Representative (LAR) for minor subject's administration of one artificial tear onto the ocular surface. A temporal view video recording will be obtained. Subjects age 11 or older will self-administer the eye drops. Subjects age 10 or younger will have eye drops administer by the subject's LAR. Adult subjects or LAR will administer the drop with their dominant hand in the eye of the subject's preference.

Subjects age 11 or older shall be in a seated position while the eye drops are self-administered. Subjects age 10 or younger can either be seated or laid based on the LAR's preference.

There will be a total of three eye drop administration attempts - two attempts on the first visit (Day 0) and one attempt at second visit (Day 30 +/- 7 days). The first eye drop administration attempt will be without coaching. The subject will then receive eye drop administration technique improvement coaching by study staff and a second eye drop administration with video recording will be obtained. One month later, the subject will return at visit 2 for a third attempt for eye drop administration without any additional coaching (to observe the retention of previous eye-drop administration technique coaching) and a video recording will be obtained.

All video recordings will then be retrospectively evaluated by independent ophthalmologist and optometrist graders according to pre-specified success and failure criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients or parents of minor patients who consent to participating in the study

Exclusion Criteria:

* Any patient who does not consent to study participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consented, routine, and real world eyecare clinic patient population, regardless of age, with or without visual impairment, willing to administer an artificial tear with video capture.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who meet pre-specified "success" criteria for proper administration of eye drop onto ocular surface on first attempt session as evaluated by the ophthalmologist or optometrist grader | There will be a total of three eye drop administration attempts - Two attempts occur on the first visit (Day 0)
  Eye drop administration success = one drop accurately falling onto the ocular surface with single drop administration without the tip of the eye drop bottle touching the hands or eye (including the eyelid, conjunctiva, eyelashes)

SECONDARY OUTCOMES:
Proportion of patients who meet each individual failure criterion on first, second, and third attempt session | three eye drop administration attempts - Two attempts on the first visit (Day 0) and one attempt at second visit (Day 30 +/- 7 days).
  Eye drop administration failure =
  * Two or more eye drops administered onto the eye
  * Eye drop missing the eye
  * Touching the tip of the eye drop bottle to the eyelid, conjunctiva, eyelashes, or hands
Proportion of patient eye drop administration "success" as evaluated by patient self-assessment on first, second, and third attempt sessions | three eye drop administration attempts - Two attempts on the first visit (Day 0) and one attempt at second visit (Day 30 +/- 7 days).
  Patient self-evaluation success = a rating of 6 or higher on Likert scale
Agreement between optometrist and ophthalmologist graders and patient eye drop administration "success" outcomes on first, second and third attempt sessions as measured by calculated Kappa statistic. | three eye drop administration attempts - Two attempts on the first visit (Day 0) and one attempt at second visit (Day 30 +/- 7 days)
  Physician evaluated eye drop administration success = one drop accurately falling onto the ocular surface on the first attempt
  • Patient self-evaluation success = a rating of 6 or higher on Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cataract Surgeons for Improved Eyecare(CSIE). Analysis of the economic impacts of dropless cataract therapy on Medicare, Medicaid, state governments, and patient costs. October 2015. http://stateofreform.com/wp-content/uploads/2015/11/CSIE_Dropless_Economic_Study.pdf
- [Result] An JA, Kasner O, Samek DA, Levesque V. Evaluation of eyedrop administration by inexperienced patients after cataract surgery. J Cataract Refract Surg. 2014 Nov;40(11):1857-61. doi: 10.1016/j.jcrs.2014.02.037. Epub 2014 Sep 22. PMID 25248295
- [Result] Hennessy AL, Katz J, Covert D, Kelly CA, Suan EP, Speicher MA, Sund NJ, Robin AL. A video study of drop instillation in both glaucoma and retina patients with visual impairment. Am J Ophthalmol. 2011 Dec;152(6):982-8. doi: 10.1016/j.ajo.2011.05.015. Epub 2011 Aug 6. PMID 21821228